CLINICAL TRIAL: NCT04753151
Title: The Study of the Effects of the Administration of Tranexamic Acid or Placebo on Perioperative Bleeding in Adults Undergoing Liver Transplantation.
Brief Title: The Effects of Tranexamic Acid or Placebo on Perioperative Bleeding in Adults Undergoing Liver Transplantation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: University of Sao Paulo (Other); Santa Casa de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 40693520.8.0000.5327
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hemorrhage
Keywords: Hemorrhage; Major bleeding; Liver transplantation; Tranexamic acid; Antifibrinolytic drugs
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized parallel controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The method for blinding the study will be carried out through the use of sealed envelopes and will include the blinding of the assisting anesthesiologists, patients, researchers, evaluators and those responsible for the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): Patients scheduled for liver transplantation and allocated for treatment with tranexamic acid (Group 1).
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Patients scheduled for liver transplantation and allocated for treatment with placebo (Group 2).
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — The study will be designed as a prospective, double-blinded clinical trial, compared to placebo (0.9% saline) in combination with conventional treatment. Patients will receive intravenous administration of 10 mg / kg tranexamic acid or placebo (0.9% saline) for 10 minutes in the 20 minutes prior to the estimated skin incision. Right after the skin incision, a maintenance dose of 1 mg / kg / h of tranexamic acid (or equivalent infusion rate of 0.9% saline) will be started, remaining until the end of the suture of the surgical wound.

SUMMARY:
Around 230 million major procedures are performed worldwide each year. Postoperative complications after major surgery, especially in solid organ transplants, are associated with a significant increase in costs and mortality. Major bleeding episodes in major surgeries such as liver transplantation are related to a significant impact on morbidity and mortality.

In this multicenter study, we aimed to compare the efficacy of tranexamic acid when compared to placebo, administered after anesthetic induction and in continuous infusion during the procedure, on the rate of intraoperative bleeding in adult patients undergoing liver transplantation. Considering its mechanism of action and its pharmacological and clinical properties, we expect to observe a significant reduction in the bleeding rate and in the need for blood components in the perioperative period of adult patients undergoing orthotopic liver transplantation.

In this study, only adult ASA III to IV patients (18 to 70 years old), scheduled for orthotopic liver transplantation at the Hospital de Clínicas de Porto Alegre, Santa Casa de Porto Alegre and at the Hospital das Clínicas of the University of Sao Paulo will be included. Exclusion criteria consider patients with a history of acute arterial thrombosis or venous thromboembolism (<1 month), patients with a history of known thrombophilia, Budd-Chiari syndrome, primary biliary cholangitis, primary sclerosing cholangitis, patients with reduced left ventricular function ( ejection fraction <40%), pulmonary hypertension, preoperative pulmonary edema, or severe preoperative hemodynamic changes requiring the use of vasoactive drugs, planned use of tranexamic acid systemically during surgery, hypersensitivity or known allergy to acid tranexamic, history of seizure disorder, patients who have recently suffered a stroke or myocardial infarction (<1 month), patients with subarachnoid hemorrhage in the last 30 days and patients previously undergoing cranial neurosurgery.

Major bleeding in this study will be defined as bleeding that results in hemoglobin ≤ 8.0 g / dL and the patient receiving a transfusion of ≥ 1 unit of red blood cells; results in a drop in hemoglobin ≥ 4.0 g / dL and the patient receives a transfusion of ≥ 1 unit of red blood cells; results in the patient receiving a transfusion of ≥ 4 units of red blood cells over a 24-hour period; or bleeding leading to surgical reintervention.

DETAILED DESCRIPTION:
In this study, only adult ASA III to IV patients (18 to 70 years old), scheduled for orthotopic liver transplantation at the Hospital de Clínicas de Porto Alegre, Santa Casa de Porto Alegre and at the Hospital das Clínicas of the Faculty of Medicine, will be included. Medicine at the University of São Paulo. All hospitals involved will be of equal importance, varying participation according to the number of liver transplant surgeries performed at the institutions. Patients with a history of acute arterial thrombosis or venous thromboembolism (<1 month), patients with a history of known thrombophilia, Budd-Chiari syndrome, primary biliary cholangitis, primary sclerosing cholangitis, patients with reduced left ventricular function ( ejection fraction <40%), pulmonary hypertension, preoperative pulmonary edema, or severe preoperative hemodynamic changes requiring the use of vasoactive drugs, planned use of tranexamic acid systemically during surgery, hypersensitivity or known allergy to acid tranexamic, history of seizure disorder, patients who have recently suffered a stroke or myocardial infarction (<1 month), patients with subarachnoid hemorrhage in the last 30 days and patients previously undergoing cranial neurosurgery. Patients with chronic dialysis kidney disease or patients in need of a liver-kidney transplant will also be excluded from the study.

To calculate the sample size, considering a 95% confidence interval and an 80% power and aiming to detect a statistical difference in the incidence of major bleeding of approximately 24% in patients in the placebo group and 14% among patients exposed to tranexamic acid, a sample of 128 patients was estimated, approximately 64 patients for each study group. The main outcome considered for the calculation of the sample size was the presence of major bleeding requiring transfusion in the perioperative period (intraoperative and in the first 24 hours postoperatively). In order to overcome possible losses during the treatment protocol, the estimated sample will be increased by approximately 10% in its final number, totaling an estimated sample of 140 patients divided into two treatment groups or arms (70 patients for each study group) .

Major bleeding in this study will be defined as bleeding that results in hemoglobin ≤ 8.0 g / dL and the patient receiving a transfusion of ≥ 1 unit of red blood cells; results in a drop in hemoglobin ≥ 4.0 g / dL and the patient receives a transfusion of ≥ 1 unit of red blood cells; results in the patient receiving a transfusion of ≥ 4 units of red blood cells over a 24-hour period; or bleeding leading to surgical reintervention.

Bleeding in the postoperative period during the hospitalization of the patient in the intensive care unit (ICU) will be assessed by the nursing staff through the flow of abdominal drains routinely used in liver transplant surgery and recorded in medical records every six hours or before bleeding. increased. In addition to bleeding, clinical, hemodynamic and laboratory / gasometric parameters will be considered for clinical or surgical intervention in the patient.

The sample calculation for this study was based on two recent previous studies. An observational study demonstrated the need for transfusion of at least one unit of packed red blood cells in approximately 24% of liver transplants and a recent systematic review demonstrated a reduction of approximately 41% in the transfusion rate of blood components related to intraoperative administration of tranexamic acid when compared to placebo in patients undergoing major non-cardiac and non-orthopedic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ASA III to IV (18 to 70 years), scheduled for orthotopic liver transplantation.

Exclusion Criteria:

* Patients with a history of acute arterial thrombosis or venous thromboembolism (<1 month), patients with a history of known thrombophilia, Budd-Chiari syndrome, primary biliary cholangitis, primary sclerosing cholangitis, patients with reduced left ventricular function (ejection fraction <40%), pulmonary hypertension, preoperative pulmonary edema, or severe preoperative hemodynamic changes requiring the use of vasoactive drugs, planned use of tranexamic acid systemically during surgery, hypersensitivity or known allergy to acid tranexamic, history of seizure disorder, patients who have recently suffered a stroke or myocardial infarction (<1 month), patients with subarachnoid hemorrhage in the last 30 days and patients previously undergoing cranial neurosurgery. Patients with chronic dialysis kidney disease or patients in need of a liver-kidney transplant will also be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative major bleeding in patients undergoing orthotopic liver transplantation. | 24 hours
  To evaluate the efficacy of tranexamic acid intravenously in relation to placebo (control - saline) on the incidence of major bleeding in the intraoperative and immediate postoperative (24 hours) in patients undergoing orthotopic liver transplantation.

SECONDARY OUTCOMES:
Effects of tranexamic acid or placebo on the mortality rate in patients undergoing orthotopic liver transplantation. | 30 days
  To evaluate the effects of tranexamic acid or placebo (control - saline) on the mortality rate (up to 30 days) in patients undergoing orthotopic liver transplantation.
Effects of tranexamic acid or placebo on the transfusion rate of blood products in the perioperative period in patients undergoing orthotopic liver transplantation. | 24 hours
  To evaluate the effects of tranexamic acid or placebo (control - saline) on the transfusion rate of blood products in the perioperative period (24 hours) in patients undergoing orthotopic liver transplantation.
Effects of tranexamic acid or placebo on the rate of fluid administration in the perioperative period in patients undergoing orthotopic liver transplantation. | 24 hours
  To evaluate the effects of tranexamic acid or placebo (control - saline) on the rate of fluid administration in the perioperative period (24 hours) in patients undergoing orthotopic liver transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Andre P Schmidt, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Andre Prato Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No